CLINICAL TRIAL: NCT03492151
Title: Confocal Laser Endomicroscopy as an IMaging Biomarker for the Diagnosis of Pancreatic Cystic Lesions
Acronym: CLIMB
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: American College of Gastroenterology (Other); The National Pancreas Foundation (Other)
Responsible Party: Principal Investigator, Somashekar Krishna, Principal Investigator, Ohio State University
Other Study IDs: 2017C0192
Record Dates: First submitted 2018-04-02; First posted 2018-04-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cyst
Keywords: Confocal laser endomicroscopy; pancreatic cancer; IPMN
MeSH Terms: conditions — Pancreatic Cyst; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Pancreas cyst fluid from EUS-nCLE
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study schema is shown in Figure 4. (A) All patients referred to one of the participating academic centers for EUS evaluation of the PCL will be enrolled in the protocol if they satisfy inclusion criteria. Patient consent will be obtained during the clinic visit or prior to their EUS. EUS-guided nCLE imaging is first performed (B) followed by EUS-guided FNA and aspiration of cyst fluid. The cyst fluid is analyzed for CEA and cytology. As per institutional standard of care, the cyst fluid is also sent for molecular analysis. The results of the cyst fluid molecular analysis (B) will be utilized for the most likely diagnosis. Based on institutional multidisciplinary tumor board meetings, surgery is performed as indicated (C). Surgical histopathology serves as "gold standard" for diagnosis. It is anticipated that the majority of patients will undergo surgical resection after their EUS.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years or older
* All patients referred for EUS-FNA of accessible PCL where surgery is contemplated
* Minimum cyst size should be ≥ 2.0 cm as determined by prior cross-sectional imaging studies

Exclusion Criteria:

* Unable to obtain informed consent
* Unable to tolerate the procedure
* Women with known pregnancy at time of procedure
* Patient age less than 18 years
* Bleeding diathesis
* Known allergy to fluorescein
* Prior pancreatic cancer
* Prior pancreatic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects for this study will be identified from patients referred for diagnostic EUS-FNA of PCLs for a non-study indication by a physician responsible for their care (i.e., gastroenterologists, oncologists, general internists, and surgeons) either at the primary study center.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of PCL diagnosis | 48 months
  Diagnostic accuracy of confocal laser endomicroscopy and/or cyst fluid molecular markers and/or composite clinical and imaging features for the diagnosis of mucinous PCLs, PCLs with malignant potential, specific PCL types, and mucinous PCLs with advanced neoplasia.
Accuracy of risk-stratification of IPMNs | 48 months
  Diagnostic accuracy of confocal laser endomicroscopy and/or composite clinical and imaging features for the risk stratification of IPMNs

SECONDARY OUTCOMES:
Imaging quality | 48 months
  Optimal quality of imaging obtained during in vivo confocal laser endomicroscopy of pancreatic cystic lesions

CONTACTS AND LOCATIONS:
Overall Officials: Somashekar Krishna, MD, MPH, Principal Investigator — Ohio State University
Locations (10):
- United States (10):
  - Mayo Clinic Scottsdale Campus, Scottsdale, Arizona
  - Stanford Hospital, Stanford, California
  - Yale School of Medicine, New Haven, Connecticut
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - NYU Langone Health, Garden City, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Firkins SA, Chen W, Krishna SG. Morphologic and Microscopic Characterization of an Unusual Pancreatic Cystic Lesion. Gastroenterology. 2021 May;160(6):e14-e16. doi: 10.1053/j.gastro.2020.09.046. Epub 2020 Oct 8. No abstract available. PMID 33039474